CLINICAL TRIAL: NCT01463995
Title: Prognosis in Neurological Intensive Care Unit Patients (proNICU Cohort)
Acronym: proNICU
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. med. Andreas Meisel, Charite University, Berlin, Germany
Other Study IDs: proNICU cohort
Record Dates: First submitted 2011-10-31; First posted 2011-11-02 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Neurological Diseases
Keywords: severe neurological diseases; neurological intensive care unit; prediction; long-term outcome; biomarkers; prediction of long-term outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (serum, plasma), cerebrovascular fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- severe neurological diseases: Patients with severe neurological diseases treated on the neurological intensive care unit

SUMMARY:
This study examines the prognostic properties of immune parameters, clinical scores, electrophysiological tests (eeg, ssep, emg, eng) and functional imaging for the prediction of functional outcome one year after treatment on a neurological intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* severe neurological disease making treatment on a neurological intensive care unit necessary
* age ≥ 18
* consent by the patient or the legal representative

Exclusion Criteria:

* participation in an interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe neurological diseases treated on a neurological intensive care unit
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2012-06; Primary Completion 2016-10-03 (Actual); Study Completion 2016-10-03 (Actual)

PRIMARY OUTCOMES:
Predictive properties of immune parameters (IL6, IL10, mHLA-DR) for functional outcome one year after symptom onset | one year after symptom onset
  To evaluate of the predictive properties of immune parameters (IL6, IL10, mHLA-DR) for functional outcome one year after symptom onset

SECONDARY OUTCOMES:
To evaluate of the predictive properties of clinical scores for functional outcome one year after symptom onset | one year after symptom onset
  To evaluate of the predictive properties of clinical scores for functional outcome one year after symptom onset
To evaluate of the predictive properties of electrophysiological measurements one year after symptom onset | one year after symptom onset
  To evaluate of the predictive properties of electrophysiological measurements one year after symptom onset
To evaluate of the predictive properties of conventional (DTI) and functional imaging (resting state) one year after symptom onset | one year after symptom onset
  To evaluate of the predictive properties of conventional (DTI) and functional imaging (resting state) one year after symptom onset
Transcriptome analyses | one year after symptom onset
  To perform transcriptome analyses to identify new biomarkers which may predict the one year- neurological outcome
Predictive properties of immune parameters in the cerebrovascular fluid for functional outcome one year after symptom onset | one year after symptom onset
  To evaluate of the predictive properties of immune parameters in the cerebrovascular fluid for functional outcome one year after symptom onset
Quality of life and occurence of depression in patients one year after symptom onset | one year after symptom onset
  To investigate the quality of life and the occurence of depression in patients one year after symptom onset
Quality of life and the occurence of depression and burnout syndrome in relatives | one year after symptom onset
  To investigate the quality of life and the occurence of depression and burnout syndrome in relatives of patients treated on the neurological intensive care unit one year after symptom onset

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, MD, Principal Investigator — Charite University Berlin (Center for Stroke Research Berlin CSB & NeuroCure Clinical Research Center NCRC)
Locations (1):
- Charite University (Center for Stroke Research Berlin CSB & NeuroCure Clinical Research Center NCRC), Berlin, Germany